CLINICAL TRIAL: NCT06616454
Title: The Effect of Time-Restricted Feeding on Body Composition and Some Metabolic Parameters in Obese Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sümeyra Başar (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor-Investigator, Sümeyra Başar, project manager, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/828
Record Dates: First submitted 2024-09-11; First posted 2024-09-27 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Adolescent Obesity
Keywords: Pediatric Obesity; Body Composition; Healthy Diet; Time-Restricted Eating
MeSH Terms: conditions — Pediatric Obesity; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: This study was planned as a randomized controlled parallel design study in 60 adolescents with obesity (BMI% ≥ 95th percentile) aged 12-18 years (between puberty stage: 5) who were followed at Erciyes University Mustafa Eraslan and Fevzi Mercan Children's Hospital. Patients will be randomized to one of two treatment groups for a 12-week intervention.
  Group 1: Intervention group - Time-restricted feeding - Ad libitum feeding between 10:00-18:00 hours
  Group 2: Control group - Calorie-restricted feeding - Nutrition plan prepared in line with the principles of the Mediterranean Diet without time restrictions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group - Calorie-restricted feeding (Experimental): Participants will be applied a nutrition plan prepared in line with the principles of the Mediterranean Diet without any time restrictions.
  Interventions: Behavioral: Intervention group - Time restricted feeding
- Intervention group - Time restricted feeding (Experimental): Participants will be applied with an ad libitum nutrition plan between 10:00 and 18:00.
  Interventions: Behavioral: Intervention group - Time restricted feeding

INTERVENTIONS:
Behavioral: Intervention group - Time restricted feeding — Participants will be applied with an ad libitum nutrition plan between 10:00-18:00.

SUMMARY:
Obesity is now recognized as a serious public health problem. It is known that obesity seen in adolescence is largely carried over to adulthood. Therefore, its treatment is important both in terms of protecting current health and preventing diseases in adulthood. Reducing energy intake plays an important role in the treatment of obesity. However, long-term adherence and effectiveness to energy restriction appear to be limited. Therefore, the need for interventions that are "effective in body weight loss" and "accessible, simple and lifestyle modification to increase dietary compliance" is clear. Time-restricted feeding is a specialized intermittent fasting protocol that includes consistent fasting and eating periods over a 24-hour cycle by supporting circadian rhythms. Especially in the adult population, positive effects of time-restricted feeding such as weight loss and blood glucose regulation are observed. However, there are limited data on this subject for adolescents. Today, the Mediterranean diet, which is one of the nutrition models that supports health, is a beneficial nutritional model that reduces body weight and obesity-related comorbidities by limiting total energy intake. However, no study has been found in the literature in which the effectiveness of time-restricted nutrition, which is a new and promising approach, and the Mediterranean diet, which is a sustainable diet model, are evaluated together. Therefore, in this study, it was aimed to evaluate the effects of planned time-restricted nutrition compatible with circadian rhythm and energy-restricted feeding planned according to the Mediterranean diet model on body composition and various metabolic parameters in obese adolescents. 60 obese adolescents aged 12-18 years will be included in this randomized controlled and parallel design study. Participants will be randomized to one of two treatment groups for a 12-week intervention. The time-restricted feeding group will form the intervention group of the study, and the energy-restricted feeding group will form the control group. Anthropometric measurements of the participants at the beginning and end of the study will be taken, and various biochemical parameters will be evaluated with the body composition and blood samples to be taken. As a result of the study, it is expected to determine the effectiveness of time-restricted feeding compared to energy-restricted feeding in terms of dietary compliance, body composition and biochemical changes.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12-18 with puberty stage:5
* Obese adolescents with a metabolic disorder (such as fatty liver, insulin resistance, prediabetes, dyslipidemia) (BMI≥95th percentile for age)
* Those who have a stable body weight for 3 months before the start of the study (current weight gain or loss <4 kg)
* Those who own and can use a Smartphone with Apple iOS or Android operating system
* Those who speak, read and understand Turkish

Exclusion Criteria:

* Those with any endocrine disorder, metabolic, chronic or major psychiatric disease other than obesity, insulin resistance, dyslipidemia, prediabetes, fatty liver
* Polycystic ovary syndrome (PCOS)
* Those with physical or mental disabilities
* Those with allergies, intolerances or eating disorders
* Those who smoke and drink alcohol
* Use of drugs that may affect study results, circadian rhythms or metabolism (such as antidiabetics, steroids, beta blockers, adrenergic stimulating agents, laxatives, etc.)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Changes in body weight | Baseline, Week 4, Week 8 and Week 12
  Changes in body weight will be examined as a result of the implemented nutrition plan.
Changes in body fat percentage | Baseline, Week 4, Week 8 and Week 12
  Changes in body fat percentage as a result of the implemented nutrition plan will be examined. The fat percentage will be assessed based on measurements taken with bioimpedance analysis devices.
Changes in body mass index | Baseline, Week 4, Week 8 and Week 12
  Changes in body mass index as a result of the implemented nutrition plan will be examined. Body mass index (BMI) will be calculated based on changes in height (cm) and weight (kg) values, using the formula kg/m².
Biochemical changes | Baseline and Week 12
  As a result of the implemented nutrition plan, changes in fasting glucose (mg/dL), total cholesterol (mg/dL), LDL cholesterol (LDL-C; mg/dL), HDL cholesterol (HDL-C; mg/dL), and triglycerides (mg/dL) levels will be evaluated.
Changes in glycated hemoglobin levels | Baseline and Week 12
  As a result of the implemented nutrition plan, changes in glycated hemoglobin (HbA1c) levels will be evaluated.
Changes in insulin levels | Baseline and Week 12
  As a result of the implemented nutrition plan, changes in insulin levels (measured in µIU/mL) will be evaluated.
Changes in hormone levels | Baseline and Week 12
  At the conclusion of the implemented nutrition plan, changes in the levels of leptin, ghrelin, adiponectin, irisin, and nesfatin hormones (ng/mL) will be evaluated.
Changes in inflammatory markers | Baseline and Week 12
  At the conclusion of the implemented nutrition plan, changes in various inflammation markers, including interleukin (IL)-17, IL-10, IL-6, IL-1β, and TNF-α (ng/mL), will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyra Başar, Study Director — sumeyra_akalin@hotmail.com
Locations (1):
- Mustafa Eraslan and Fevzi Mercan Children's Hospital, Kayseri, Turkey (Türkiye)